CLINICAL TRIAL: NCT06324279
Title: The Cervical Sliding Sign as a Marker in Prediction of Successful Induction of Labor
Brief Title: Cervical Sliding Sign to Predict Outcome of Induction of Labor
Status: Active, not recruiting | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Omaima Abbas Mahmoud, Resident, Ain Shams Maternity Hospital
Other Study IDs: 000017585
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Induction of Labor; Transvaginal Ultrasound: Cervical Sliding Sign
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- term pregnant women with Singleton living fetus attending for induction of labor
  Interventions: Device: Transvaginal ultrasound; Drug: Misoprostol 200mcg Tab

INTERVENTIONS:
Device: Transvaginal ultrasound — Transvaginal ultrasound will be used to see the presence of cervical sliding sign
Drug: Misoprostol 200mcg Tab — Induction of labor by misoprostol

SUMMARY:
Assess the role of transvaginal ultrasound specifically a sign called cervical sliding sign, in the prediction of success of induction of labor.

The prediction of outcome of induction of labor has always been an important topic to all obstetricians. Bishop score is traditionally considered reliable way to predict the outcome of induction of labor by assessing the cervical dilatation, effacement, position, and consistence and assessing the level of the fetal head in the birth canal. Since The bishop score remains a highly subjective method for prediction of outcome of induction of labor, the use of sonographic measurements such as cervical sliding sign can be a better predictor of successful induction of labor.The presence of CSS was defined as the sliding of the anterior cervical lip on the posterior one under gentle pressure of the transvaginal probe.

Patients undergoing induction of labor with misoprostol will be checked for the cervical sliding sign. The mode of delivery, induction to active labor time and active labor to delivery time will be recorded and analysed to assess whether the sliding sign is an independent predictor of success of induction.

DETAILED DESCRIPTION:
Induction of labor is a common practice in modern obstetrics. It is the use of mechanical or pharmacological -or both ways- to stimulate uterine contractions before spontaneous labor to induce cervical dilatation and delivery. Induction of labor at term have many advantages. It can reduce to risk of still birth. It also reduces the risk of macrosomia and its adverse outcomes such as maternal trauma, shoulder dystocia or the need for instrumental delivery (Kim, et al., 2019). However, induction of labor can also have adverse outcomes, the most common is failure and increasing the risk of cesarean section. Induction of labor may not be tolerated by some patients because of the potential increase in the duration of labor or a prolonged latent phase. Increased cost compared to spontaneous delivery course and possible neonatal morbidity if the gestational age is less than 39 weeks of gestation are other drawbacks. (Kim, et al., 2019) Since the success of induction of labor is related to the condition of the cervix, investigators have proposed the importance of having a reliable system for determining the cervical maturity. A number of studies considered the use of sonographic measurement of cervical length to predict the success of labor induction. The sonographic marker for assessing the cervical softening called the cervical sliding sign (CSS) which was introduced by (Volpe, et al., 2019), demonstrated its correlation with the occurrence of impending delivery in women with preterm uterine contractions. The performance of the CSS in predicting the success of IOL was conducted in two academic centers by (Volpe, et al., 2022). However, its generalizability to community hospitals cannot be certain and needs further testing. The presence of CSS was defined as the sliding of the anterior cervical lip on the posterior one under gentle pressure of the transvaginal probe. (Volpe, et al., 2022)

Aim/ Objectives. Assess the role of the cervical sliding sign (CSS) as a marker in the prediction of the outcome of induction of labor (IOL) at term gestation.

Research Hypothesis:

The presence of Cervical Sliding sign in pregnant women at term gestation planned for Induction of labor predicts a higher chance of vaginal delivery within 24 hours.

Research Question:

Is CSS a successful marker for prediction of outcome of induction of labor in pregnant women at term gestation? Methodology

Type of Study: Prospective observational cohort study Study Setting: Ain Shams University Maternity Hospital (labor ward). Study period: 6 months Study Population: The study will be conducted on term pregnant women with Singleton living fetus attending Ain Shams University Maternity Hospital for induction of labor with the following criteria:

Inclusion criteria:

1. women age: from 18 to 35 years old.
2. Single living term fetus with gestational age ≥ 37 weeks. 3- Eligible for IOL. 4- Bishop score <6 5- Estimated fetal weight < 4Kg.

Exclusion criteria:

1. previous caesarean section. (increases risk of rupture uterus)
2. Multiple pregnancy, IUFD, preterm or macrosomic fetus (defined as fetus >4.5kg or fetus of diabetic mother >4Kg) (increases risk of shoulder dystocia)
3. Women with major uterine anomalies. (appendix A: ESHRE/ESGE classification for Female genital tract anomalies (Grimbizis GF, et al,. 2013) (increases risk of CS)
4. Vasa previa, placenta previa (increases risk of antepartum hemorrhage)
5. previous myomectomy reaching the endometrial cavity. (Increases risk of rupture uterus)

7- patient refuse to participate or inability to consent. (patient's right to refuse).

Sample Size and sample Size Justification:

Using the PASS 15 program for sample size calculation, reviewing results from a previous study (Volpe et al.2022) showed that the cervical sliding sign (CSS) was found in 48% of the study group (non-consecutive series of uncomplicated singleton term pregnancies, planned for IOL, with a fetus in cephalic presentation patients), based on this frequency and after 20% adjustment for dropout rate, a sample size of at least 130 participants produces a two-sided 95% confidence interval with a width equal to 0.199 when the sample proportion is 0.480.

Ethical Consideration:

This study will be done after approval of the ethical committee of the department of obstetrics and gynecology, faculty of medicine, Ain Shams University. Informed consent will be taken from all participants before recruitment in the study, and after explaining the purpose and procedures of the study. The investigator will obtain the written, signed informed consent of each subject prior to performing any study specific procedures on the subject. The investigator will retain the original signed informed consent form. All laboratory specimens, evaluation forms, reports, video recordings and other records that leave the site will not include unique personal to maintain subject confidentiality. The study will be based on the investigator self-funding.

Study procedures and interventions:

Women fitting into our inclusion criteria will be subjected to:

1. history taking (personal, obstetric, medical and surgical)
2. Transvaginal ultrasound to assess the presence of CSS with a semi-filled bladder using a 10 MHz endo-vaginal probe EC3-10T of Alpinion E-CUBE 5 ultrasound machine (ALPINION MEDICAL SYSTEMS Co., Ltd. Guro-gu, Seoul, 08393, Republic of Korea) will be done by the most senior resident. "The CSS will be evaluated as follows:

1- acquisition of a sagittal view of the cervix, on which the internal and external os and the endocervical canal could be identified. 2- Gentle pressure with the transvaginal probe on the cervix until maximum compression of the cervix is achieved. 3- Visualization of the anterior cervical lip "sliding" on the posterior one is defined as the presence of CSS." (Volpe, et al., 2022) 3- Induction and management of labor will be conducted following the hospital's protocol (APPENDEX B: FIGO MISOPROSTOL-ONLY RECOMMENDED REGIMENS 2017(Morris JL, et al., 2017)) 4- record the mode of delivery for each participant either vaginal delivery or cesarean deliveries. 5- Measurement of induction-to-active-labor1 time (active labor time defined as ≥ 6cm dilated cervix), active-labor-to-delivery time, total length of labor.

Outcomes:

* 1ry outcome: successful vaginal delivery.
* 2ry outcomes:

  * induction-to-active-labor time interval.
  * Active -labor-to-delivery time interval.
  * Mode of Delivery (vaginal/ Instrumental/ Cesarean)
  * Reason for CS (Fetal distress/ failure of induction/ failure of progress).

Statistical analysis:

- All data will be collected, tabulated, and statistically analyzed by software package program

ELIGIBILITY:
Inclusion Criteria:

* 1. women age: from 18 to 45 years old.

  2. Single living term fetus with gestational age ≥ 37 weeks.

  3- Eligible for IOL. 4- Bishop score <6 5- Estimated fetal weight < 4Kg.

Exclusion Criteria:

* 1- previous caesarean section. (increases risk of rupture uterus) 2- Multiple pregnancy, IUFD, preterm or macrosomic fetus (defined as fetus

>4.5kg or fetus of diabetic mother >4Kg) (increases risk of shoulder dystocia) 3- Women with major uterine anomalies. (appendix A: ESHRE/ESGE classification for Female genital tract anomalies (Grimbizis GF, et al,. 2013) (increases risk of CS) 4- Vasa previa, placenta previa (increases risk of antepartum hemorrhage) 5- previous myomectomy reaching the endometrial cavity. (Increases risk of rupture uterus) 7- patient refuse to participate or inability to consent. (patient's right to refuse).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will be conducted on term pregnant women with Singleton living fetus attending Ain Shams University Maternity Hospital for induction of labor
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Mode of delivery | 48 hours
  Vaginal or cesarean section
Induction to active labor time | 48 hours
  Start of induction till cervical dilation of 6 cm
Active labor to delivery time | 10 hours
  From cervical dilation of 6 cm till delivery of fetus

CONTACTS AND LOCATIONS:
Overall Officials: Omaima A Mahmoud, mbchb, Principal Investigator — Ainshams university faculty of medicine
Locations (1):
- Maternity hospital, ainshams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided